CLINICAL TRIAL: NCT02633111
Title: DNA Sequencing-Based Monitoring of Minimal Residual Disease to Predict Clinical Relapse in Aggressive B-cell Non-Hodgkin Lymphomas
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Mayo Clinic (Other); M.D. Anderson Cancer Center (Other); University of Pennsylvania (Other); University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: 15-180
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: B-cell Non-Hodgkin Lymphoma; Aggressive
Keywords: DNA Sequencing; 15-180
MeSH Terms: conditions — Lymphoma, B-Cell; Aggression | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (1):
- Patients with aggressive B-cell Non-Hodgkin lymphoma: This is a non-therapeutic protocol aimed to assess the ability of Adaptive clonoSEQ® MRD assay to detect clinical relapse in DLBCLwhen compared to conventional approaches for detecting relapse such as patient-reported symptoms, clinical exams, and CT scans.
  Interventions: Other: collected at pre-treatment tumor biopsy; Other: Peripheral blood tests; Device: PET/CT

INTERVENTIONS:
Other: collected at pre-treatment tumor biopsy — to identify the tumor-specific clonotype
Other: Peripheral blood tests — for MRD analysis at 3, 6, 9, 12, 15, 18, 21, and at relapse (+/- 1 month).
Device: PET/CT — at 3, 6, 9, 15, 18, 21 and at relapse(+/- 1 month)

SUMMARY:
The purpose of this study is to determine whether a blood test can accurately detect whether if the participant's lymphoma has come back after completion of initial chemotherapy treatment for their aggressive B-cell Non-Hodgkin lymphoma. The purpose of the study is to see if MRD in blood samples can potentially replace CT scans after completion of chemotherapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at time of signing informed consent
* Histology-confirmed aggressive B-cell Non-Hodgkin lymphoma

  * De novo diffuse large B-cell lymphoma (including all subtypes such as primary mediastinal B-cell lymphoma and T-cell rich B-cell lymphoma). According to the 2008 WHO Classification of Hematopoietic and Lymphoid Tumors. These would include double or triple-hit diffuse large B-cell lymphomas with MYC/BCL2 and/or BCL6 gene rearrangements. These cases may be classified as high grade B-cell lymphomas according to the 2017 revision of the WHO Classification of Hematopoietic and Lymphoid Tumors.
* Recipient of frontline multi-agent chemotherapy (for example, RCHOP, dose adjusted-REPOCH, RCHOP/RICE, RCHOP+investigational agent, etc). Eligible patients will have recently received (≤ 4 months from end of treatment assessment), be actively receiving, or planned to receive frontline chemotherapy in near future (within 3 months of signing consent). A frontline therapy program can include different sequential phases of treatment, including high-dose therapy and autologous stem cell transplantation.
* Required pre-treatment test specimen from bone marrow, blood, lymph node, or alternate site to identify tumor-specific clonotype.
* Ability to adhere to the study visit schedule and all the protocol requirements, including surveillance imaging and MRD test specimen collection at specified time points.

Exclusion Criteria:

* Patients receiving 2nd or greater line of therapy.
* Stage I or II disease.
* Primary mediastinal B-cell lymphoma.
* Transformation from antecedent or coincident indolent B-cell Non-Hodgkin lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
MRD assay to predict clinical relapse | 2 years
  using the Sequenta diagnostic tool prior to detection using the conventional means (clinical exams and scans) in DLBCL patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kumar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - University of Miami, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/